CLINICAL TRIAL: NCT00000951
Title: A Phase IV Randomized Study of the Use of Fluconazole as Chronic Suppressive Therapy Versus Episodic Therapy in HIV Positive Subjects With Recurrent Oropharyngeal Candidiasis
Brief Title: A Study to Compare the Use of Fluconazole as Continuous Therapy Versus Periodic Therapy in HIV-Positive Patients With Recurrent Thrush
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 323; 11297 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Candidiasis, Oral; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Fluconazole; Antifungal Agents; Candidiasis, Oral; Drug Administration Schedule; Pharyngeal Diseases
MeSH Terms: conditions — Candidiasis, Oral; HIV Infections; AIDS-Related Opportunistic Infections; Pharyngeal Diseases | interventions — Fluconazole

INTERVENTIONS:
Drug: Fluconazole

SUMMARY:
The purpose of this study is to determine whether it is better to treat patients with fluconazole on a continuous basis to prevent thrush (yeast infection in the mouth) from coming back or to wait and treat each episode of thrush.

Fluconazole is one of the most commonly prescribed drugs to treat thrush and other yeast infections. However, the number of patients with fluconazole-resistant thrush is increasing, and it is not known whether continuous or intermittent use of fluconazole leads to greater resistance. Therefore, it is important to determine the most effective treatment strategy.

DETAILED DESCRIPTION:
This study will evaluate two different management strategies for patients with advanced HIV infection who are at risk for recurrent and fluconazole-refractory oropharyngeal candidiasis. The treatment duration will be at least 24 months in order to evaluate the long-term effects of the treatment strategies on the development of fluconazole-refractory thrush. In addition to investigating antifungal treatment as it relates to fluconazole-refractory infections, the study will evaluate host factors and organism-related factors in order to increase our understanding of the pathogenesis of oropharyngeal candidiasis and fluconazole-refractory infections.

Prior to randomization to a long-term management strategy using fluconazole, patients are stratified into one of three groups according to their baseline CD4+ count (cells/mm3): 0-49, 50-100, and 101-150. Patients without oropharyngeal candidiasis (no thrush present) at enrollment and those patients who respond (no thrush present) to the initial acute therapy for an active infection are randomized 1:1 to one of two management strategies for fluconazole: Arm A (episodic therapy) or Arm B (chronic suppressive therapy with continuous fluconazole). Patients are then followed for a duration of 24 months after enrollment of the last subject. Patients with active oropharyngeal candidiasis at time of enrollment will be treated with fluconazole for up to 2 weeks and patients who respond (no thrush present) are then randomized to a long-term management strategy. Those who do not respond (refractory disease) to the acute treatment are permanently discontinued from the study. Women in both groups will have the option of being treated for vulvovaginal candidiasis either through or outside the study.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Have a CD4+ cell count less than 150 cells/mm3.
* Had at least one episode of thrush in the 24 months before study entry.
* Have a life expectancy of at least 12 months.
* Weigh at least 88 pounds.
* Are 13 years of age or older (consent of parent or guardian required if under 18).
* Agree to practice abstinence or use effective methods of birth control during the study.

Exclusion Criteria

You will not be eligible for this study if you:

* Have an allergy to azoles.
* Have had 3 episodes or more of thrush within 12 weeks of study entry.
* Have a history of esophageal candidiasis.
* Have a history of fluconazole-resistant infection.
* Have an active opportunistic infection requiring treatment within 14 days before study entry.
* Have a fungal infection requiring certain medications.
* Have a severe liver disease (e.g., cirrhosis).
* Are unable to tolerate oral medications.
* Take certain medications.
* Are pregnant or breast-feeding.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 948
Dates: Study Completion 2002-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Goldman, Study Chair; Scott G. Filler, Study Chair
Locations (54):
- United States (53):
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - San Francisco Gen Hosp, San Francisco, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Howard Univ, Washington D.C., District of Columbia
  - Institute for Clinical Research, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Emory Univ, Atlanta, Georgia
  - Emory Hemo Comp Evaluation Clinic / East TN Comp Hemo Ctr, Atlanta, Georgia
  - Queens Med Ctr, Honolulu, Hawaii
  - Univ of Hawaii, Honolulu, Hawaii
  - Northwestern Univ Med School, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Louis A Weiss Memorial Hosp, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Division of Inf Diseases/ Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana / Life Care Clinic, Indianapolis, Indiana
  - Univ of Iowa Hosp and Clinic, Iowa City, Iowa
  - State of MD Div of Corrections / Johns Hopkins Univ Hosp, Baltimore, Maryland
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Boston Med Ctr, Boston, Massachusetts
  - Hennepin County Med Clinic, Minneapolis, Minnesota
  - Univ of Minnesota, Minneapolis, Minnesota
  - St Paul Ramsey Med Ctr, Saint Paul, Minnesota
  - St Louis Regional Hosp / St Louis Regional Med Ctr, St Louis, Missouri
  - Univ of Nebraska Med Ctr, Omaha, Nebraska
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Saint Clare's Hosp and Health Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - St Vincent's Hosp / Mem Sloan-Kettering Cancer Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - St Mary's Hosp (Univ of Rochester/Infectious Diseases), Rochester, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Univ of Kentucky Lexington, Cincinnati, Ohio
  - Case Western Reserve Univ, Cleveland, Ohio
  - MetroHealth Med Ctr, Cleveland, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Philadelphia Veterans Administration Med Ctr, Philadelphia, Pennsylvania
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Tennessee / E Tennessee Comprehensive Hemophilia Ctr, Knoxville, Tennessee
  - Univ of Texas Galveston, Galveston, Texas
  - Univ of Washington, Seattle, Washington
- Univ of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Background] Swindells S, Evans S, Zackin R, Goldman M, Haubrich R, Filler SG, Balfour HH Jr; AIDS Clinical Trial Group 722 Study Team. Predictive value of HIV-1 viral load on risk for opportunistic infection. J Acquir Immune Defic Syndr. 2002 Jun 1;30(2):154-8. doi: 10.1097/00042560-200206010-00003. PMID 12045677